CLINICAL TRIAL: NCT04938349
Title: Neuromechanisms of Falls in Older Adults With MCI: Targeting Assessment and Training of Reactive Balance Control
Brief Title: Dual Task Perturbation Training for OAwMCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Roybal Predoctoral pilot grant (Unknown)
Responsible Party: Principal Investigator, Tanvi Bhatt, Associate Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0478; R01AG073152 (NIH)
Record Dates: First submitted 2021-06-11; First posted 2021-06-24 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Mild Cognitive Impairment; Old Age; Debility
Keywords: Dual-task training; Mild cognitive impairment; Perturbation-based training; treadmill training; cognitive-motor training; perturbation
MeSH Terms: conditions — Cognitive Dysfunction; Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Single session dual task perturbation training-OAwMCI (Experimental): Participants will receive single session training of dual task. Six cognitive games that target working memory, executive functioning, visuomotor reactions, and language fluency will be provided in standing to get themselves familiarized. Following the cognitive tasks, participants will receive 12 slips without performing cognitive task (Single task training) at the highest intensity. Subsequently, 12 slips during standing while performing a cognitive task (dual task) will be administered. Similarly, they will then undergo 12 dual task walking trials (at self-selected speed) followed by 12 walking slips.
  Interventions: Behavioral: Dual task perturbation training
- Multiple session dual task perturbation training-OAwMCI (Experimental): All participants will undergo stance and walking perturbation training for 4 weeks. Six cognitive games that target working memory, executive functioning, visuomotor reactions, and language fluency will be provided in standing to get themselves familiarized. Following the cognitive tasks, participants will receive 12 slips without performing cognitive task (Single task training) at the highest intensity. Subsequently, 12 slips during standing while performing a cognitive task (dual task) will be administered. Similarly, they will then undergo 12 dual task walking trials (at self-selected speed) followed by 12 walking slips.
  Interventions: Behavioral: Dual task perturbation training
- Single session dual task perturbation training-CIOA (Active Comparator): All participants will receive only one training session of dual task. Six cognitive games that target working memory, executive functioning, visuomotor reactions, and language fluency will be provided in standing to get themselves familiarized. Following the cognitive tasks, participants will receive 12 slips without performing cognitive task (Single task training) at the highest intensity. Subsequently, 12 slips during standing while performing a cognitive task (dual task) will be administered. Similarly, they will then undergo 12 dual task walking trials (at self-selected speed) followed by 12 walking slips.
  Interventions: Behavioral: Dual task perturbation training

INTERVENTIONS:
Behavioral: Dual task perturbation training — Participants will play six cognitive games targeting working memory, executive functioning, visuomotor reactions, and language fluency provided in standing. Following which they will receive 12 slips without performing cognitive task (Single task training) at the highest intensity and 12 slips during standing while performing a cognitive task (dual task). Also, they will then undergo 12 dual task walking trials (at self-selected speed) followed by 12 walking slips.

SUMMARY:
Studies have determined that compared to cognitively intact older adults (CIOA), older adults with mild cognitive impairment (OAwMCI) exhibit more pronounced balance and gait impairments which lead to an increased risk of falls and mobility decline. Such impairments are evident during dual-tasking (i.e., simultaneous performance of cognitive and motor task) and OAwMCI have demonstrated an increased cognitive-motor interference (deteriorated performance of either or both cognitive/motor task). Furthermore, our preliminary laboratory findings indicate that compared to CIOA, OAwMCI in response to large-magnitude treadmill perturbations exhibits poor reactive responses (first line of defense against balance loss) and are unable to modulate their responses as the magnitude of perturbation increases. Despite that conventional exercise methods offer beneficial effects; they comprise of self-initiated task-specific exercises and may not focus on training reactive responses. Additionally, due to the presence of subtle balance and gait deficits, clinical measures used may not be sensitive enough to determine the risk of fall post-training. Furthermore, these training methods incorporate multiple sessions due to which adherence to exercise training is difficult with only a fraction of the older adults benefiting from it. Therefore, it is essential to incorporate a task-specific strategy that promotes factors associated with falling like balance control, muscular responses, coordination of limbs, and cognition through which OAwMCI may acquire maximum benefits to prevent a balance loss. One feasible method, which harnesses technology that can be used to deliver balance disturbances either while standing or walking in a consistent and controlled manner, is via a custom-based motorized treadmill. The scientific rigor from preliminary studies has reported a successful reduction of falls through a single session exposing CIOA to multiple treadmill-induced perturbations during gait and has shown significant improvement in reactive responses. For that reason, this stage 1 pilot study will examine the feasibility, applicability, and tolerability of a combined cognitive, and perturbation training on biomechanical determinants associated with falls and promote physical activity: kinematic variables, muscular responses, and cognitive function.

DETAILED DESCRIPTION:
Given the cognitive decline and poor reactive responses among OAwMCI, it is essential to incorporate a strategy to enhance cognition and motor performance for promoting healthy aging. For this reason, we propose this study that aims to determine the feasibility, applicability and tolerability of a dual-task perturbation training paradigm in OAwMCI. This involves a treadmill induced perturbation training while concurrently performing a cognitive task with an aim to improve effective compensatory stepping strategies to prevent balance loss. Further, while testing on laboratory induced perturbations may provide an insight into understanding kinematic variables, evaluating the change on performance-based outcome measure may be clinically useful. The overall aim of this proposal to examine the central mechanisms of reactive balance control and perturbation-training adaptation to improve fall-resisting skills in healthy older adults and people with MCI using the following set of aims. Aim 1: To examine biomechanical and neuromuscular differences during reactive balance control against mechanical perturbations during stance and gait between OAwMCI and CIOA. Compared to CIOA, OAwMCI will show: H1.1. greater falls due to impaired biomechanical (delayed step initiation, lower reactive stability and greater limb support descent) and neuromuscular responses (longer postural response latencies and fewer muscle synergies with different structural activation) on novel stance and gait perturbations, which will worsen with dual task performance; H1.2. reduced modulation (scaling) of biomechanical and neuromuscular responses with increasing perturbation intensity; H1.3. slower rate of adaptation in stability control and muscle synergy adjustment with repeated perturbation exposure.

Aim 2: To relate impairments observed during reactive balance control in perturbed stance and gait with structural brain integrity, cognition and falls in OAwMCI. These older adults will display H2.1: Lower gray matter volume in fronto-pareital cortex and brainstem, and lower white matter integrity in sensorimotor pathways which will significantly correlate with poor performance on reactive stepping response; H2.2: Lower scores on neuropsychological battery test and NIH cognitive toolbox examining domains of executive function (attention, cognitive flexibility and response inhibition), visuo-spatial awareness, episodic memory which will correlate with deteriorated reactive stepping response. H2.3: Fall-Index computed from measures of reactive stability and limb support that are obtained from perturbation-based reactive measures will better discriminate prospective laboratory induced and real-life falls than conventional instrumented (postural sway and limits of stability) and performance-based clinical measures of balance and mobility, with increased predictive accuracy of Fall-Index under dual-task conditions.

Aim 2: To determine if deficits in reactive balance responses contribute to increased falls in OAwMCI during static and dynamic tasks than CIOA especially under dual-tasking. H2.1: Measures of reactive stability and limb support under dual-task conditions during perturbed gait will best discriminate retrospective and laboratory induced falls in this population. H2.2 Predictive accuracy of Fall-Index which will be greater than of clinical measures of balance and mobility.

Aim 3: To examine the feasibility and potential effectiveness of novel 6-week perturbation-based cognitive-motor intervention for improving fall-resisting skills during perturbed stance and gait. H3.1: Post-training OAwMCI will improve stability control, cognition and reduced laboratory falls, especially under dual-task conditions. H3.2: Baseline cognition and structural brain integrity/connectivity will predict change in stability control and fall-risk. H3.3. Improvements in stability control, cognition and falls reduction will be retained for at least 3 months post withdrawal of intervention resulting in improved community ambulation and reduced fear of falling and perceived cognitive load on activities of daily living

ELIGIBILITY:
Inclusion Criteria:

* Age group: Older adults between the age group > 55 years old with MOCA less than 26 out of 30 will be classified as mild cognitive impairment and those above 26 out of 30 as cognitively intact older adults .
* Absence of any acute or chronic neurological (Stroke, Parkinson's disease, Alzheimer's disease), cardiopulmonary, musculoskeletal, or systemic diagnosis.
* No recent major surgery (< 6 months) or hospitalization (< 3 months)
* Not on any sedative drugs
* Can understand and communicate in English
* Ability to walk more than 10 meters without an assistive device

Exclusion Criteria:

* Participants will not proceed with the study if any of the following occurs at baseline measurement: 1) HR > 85% of age-predicted maximal heart rate (HRmax) (HRmax = 220 - age), 2) systolic blood pressure (SBP) > 165 mmHg and/or diastolic blood pressure (DBP) > 110 mmHg during resting), and/or 3) oxygen saturation (measured by pulse oximeter) during resting < 90%.
* History of bone fracture or significant other systemic disease or surgery in the last six months
* Specific to MRI participants: Self-reported presence of a pacemaker, metal implants other than orthopedic implants, and/or Claustrophobia, cataract surgery (lens not compatible to the MRI confirmed by the MRI technician)
* Weighs > 220 lbs (Harness weight threshold)

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2021-09-14 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Stability gain or loss | Baseline (1st novel slip, trip week 1), immediate post-training (repeated perturbation training session, week 1) and 4 weeks of training
  Stability is defined by both the position of a person's center-of-mass (COM) with respect to his or her base-of-support (BOS) and it's velocity.
Change in Limb support gain or loss | Baseline (1st novel slip, trip week 1), immediate post-training (repeated perturbation training session, week 1) and 4 weeks of training
  The inability to provide timely limb support due to insufficient amount of upward impulse generated from the ground reactive force can cause limb collapse, as characterized by the quotient of amount and rate of hip descent (Vhip/Zhip) measured from hip height and lead to an eventual fall.
Change in laboratory-induced falls | Baseline (1st novel slip, trip week 1), immediate post-training (repeated perturbation training session, week 1) and 4 weeks of training
  Perturbation is induced successfully and safely to reproduce inadvertent falls in a protective laboratory environment. Falls will be measured by the amount of body weight supported by the full-body harness system and measured by a load cell attached to this system. Instability of the body's COM and poor limb support prior to touchdown of the recovery step account for 90~100% of subsequent falls (occurring ~500ms later) in both sit-to-stand-slip and in gait-slip, in the laboratory settings. Intervention consists of repeated perturbation training to induce a change in the laboratory induced falls immediately post-training and examine it's retention after the initial training session.
Change in postural stability during reactive balance control (single and dual-task) on treadmill slips | Baseline (1st novel slip, trip week 1), immediate post-training (repeated perturbation training session, week 1) and 4 weeks of training
  Reactive balance control will be examined via the stance perturbation test under single and dual-task conditions (simultaneous performance of Letter number sequencing task or auditory stroop task). Postural stability can be defined as simultaneous control of center of mass (COM) position and velocity during slip-like or trip like perturbation relative to the rear edge of base of support (rear heel). The position is normalized with the individual's foot length, and velocity by square root of gravitational acceleration and individual's body height. Larger values indicate greater stability.
Change in postural stability during reactive balance control (single and dual-task) on overground slips | Baseline (1st novel slip, trip week 1), immediate post-training (repeated perturbation training session, week 1) and 4 weeks of training
  Reactive balance control will be examined via the stance perturbation test under single and dual-task conditions (simultaneous performance of Letter number sequencing task or auditory stroop task). Postural stability can be defined as simultaneous control of center of mass (COM) position and velocity during slip-like or trip like perturbation relative to the rear edge of base of support (rear heel). The position is normalized with the individual's foot length, and velocity by square root of gravitational acceleration and individual's body height. Larger values indicate greater stability.
Change in walking step length | Baseline (1st novel slip, trip week 1), immediate post-training (repeated perturbation training session, week 1) and 4 weeks of training
  Step length will be determined during single and dual-task walking performance via the walking on the treadmill and the GaitRite mat. Higher values for step length indicate better performance.
Change in walking cadence | Baseline (1st novel slip, trip week 1), immediate post-training (repeated perturbation training session, week 1) and 4 weeks of training
  Cadence will be determined during single and dual-task walking performance via the walking on the treadmill and the GaitRite mat. Lower cadence indicate better performance.
Change in walking stride length | Baseline (1st novel slip, trip week 1), immediate post-training (repeated perturbation training session, week 1) and 4 weeks of training
  Stride length will be determined during single and dual-task walking performance via the walking on the treadmill and the GaitRite mat. Higher values for stride length indicate better performance.
Change of accuracy in letter number sequencing | Baseline (1st novel slip, trip week 1), immediate post-training (repeated perturbation training session, week 1) and 4 weeks of training
  This is an oral trail making test which includes listing alternate letter and number from the cue given in sequence. This test will be performed under single and dual-task conditions. Higher scores indicate better performance.
Change in accuracy of Visual clock test | Baseline (1st novel slip, trip week 1), immediate post-training (repeated perturbation training session, week 1) and 4 weeks of training
  This test involves responding to the location of the minute and hour hand on a clock. This test will be performed under single and dual-task conditions. Higher scores indicate better performance.
Change in dual-task cost | Baseline (week 1), immediate post-training (repeated perturbation training session, week 1) and 4 weeks of training
  Dual-task motor and cognitive cost will be calculated using the formula- [(Dual-task performance- Single Task performance)/Single task performance]. This will be calculated for dual-task performance during intentional postural sway, reactive balance control and gait conditions. Lower cost indicates better performance.
Change in visuomotor task | Baseline (week 1), immediate post-training (repeated perturbation training session, week 1) and 4 weeks of training
  This test involves continuous tracking of a cyclic moving target on the screen using a motion sensor placed on the head. Higher scores indicates poor performance.
Fractional anisotropy | Baseline (week 1)
  White matter integrity tested using magnetic resonance imaging
Gray matter volume | Baseline (week 1)
  Gray matter volume tested using magnetic resonance imaging
Functional connectivity Z score | Baseline (week 1)
  Resting state functional connectivity using magnetic resonance imaging

SECONDARY OUTCOMES:
Perceived task load | Baseline (1st novel slip, trip week 1), immediate post-training (repeated perturbation training session, week 1) and 4 weeks of training
  NASA TLX visual analog scale will be used to determine the perceived task load after every trial is completed. Higher scores indicates poor performance.
Balance evaluation Systems test | Baseline (week 1) and 4 weeks of training
  consists of 36 different performances which will be used to determine different balance control domains such as self-initiated performances and reactive balance control, and gait functions. Each item in the scale ranges from 0 to 3 indicating severe impairment to no impairment amounting to a total score of 108 converted to percentage. Higher scores indicate better performance.
Berg Balance scale | Baseline (week 1) and 4 weeks of training
  Assess static and dynamic balance. This scale consists of the participant transferring from one chair to another, reaching forward, stepping up and down from a stepping stool, standing with eyes closed and open, one leg standing. It is a 14-item scale with each item score ranging from 0-4. Performance on the scale will be calculated on a total of 56. Less than 45 will indicate greater risk of falling.
Cognitive Timed up and Go test | Baseline (week 1) and 4 weeks of training
  Time taken to walk 3 meters as quickly as possible while concurrently performing a counting backward task. Higher scores indicate poor performance.
Muscle Strength | Baseline (week 1) and 4 weeks of training
  The isokinetic dynamometer for determining lower extremity (hip, knee, and ankle) muscle strength bilaterally. Muscle strength will be measured via Newton, i.e., force applied to perform the movement pre training compared to post training. Higher values indicate higher muscle strength.
Range of Motion | Baseline (week 1) and 4 weeks of training
  The electronic goniometer to determine range of motion of both lower extremities (hip, knee, and ankle) will be used. Range of motion will be noted in degrees and higher values indicate higher muscle strength.
Fukuda step test | Baseline (week 1) and 4 weeks of training
  Participant is asked to march (50 to 100 steps) in place with eyes closed and arms extended to 90° angle in front of the body. After completing 50 steps, if the body is rotated more than 30° angle will indicate vestibular weakness to the side rotated. Similarly, after performing 100 steps, an angle greater than 45° will indicate unilateral vestibular weakness of the side to which the body is rotated.
Head thrust test | Baseline (week 1) and 4 weeks of training
  Examiner rotates subjects head 15-30 degrees from the center and then rapidly rotates to the other side while asking the participant to look at examiner's eyes. If any nystagmus (oscillation of eyeballs horizontally or vertically) is noticed, it will indicate vestibular weakness.
Postural Sway | Baseline (week 1) and 4 weeks of training
  This test quantitatively assesses the participant's ability to use visual, proprioceptive, and vestibular inputs for maintaining their posture in quiet standing. The test will be administered under single and dual-task (simultaneous performance of motor and cognitive tasks) conditions.
Change in physical activity level (Questionnaires) | Baseline (week 1) and 4 weeks of training
  Questionnaires such as Physical Activity Scale for elderly and activity specific balance confidence scale will be self-reported by the participant. Activity specific balance confidence scale consists of 16 items, and each item score ranges from 0-100. The total score with 0 confidence indicates no confidence and 100 with complete confidence.

CONTACTS AND LOCATIONS:
Overall Officials: Tanvi Bhatt, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No